CLINICAL TRIAL: NCT00854672
Title: Exercise Capacity, Muscle Strength and Fatigue in Sarcoidosis: a Two-year Follow-up Study
Brief Title: Muscle Strength and Exercise Capacity in Sarcoidosis Patients
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ild care foundation (Other)
Responsible Party: Principal Investigator, marjolein drent, Prof. Marjolein Drent, Maastricht University Medical Center
Other Study IDs: MEC 09-4-007
Record Dates: First submitted 2009-02-26; First posted 2009-03-03 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Sarcoidosis
Keywords: Sarcoidosis; muscle strength; exercise intolerance; QOL
MeSH Terms: conditions — Sarcoidosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- sarcoidosis patients: Sarcoidosis patients referred to the ild care team of the outpatient clinic of the department of Respiratory Medicine of the MUMC and also participated in the baseline study between November 2008 and September 2009 will be included in this study

SUMMARY:
The aim of this study is to examine exercise capacity, muscle strength and fatigue in sarcoidosis. In this longitudinal study the changes in prevalence of exercise intolerance, reduced muscle strength and fatigue will be established in a two-year follow-up. Also the relation between these physical impairments in time and other clinical parameters, such as QOL, will be established.

DETAILED DESCRIPTION:
The aim of this study is to examine exercise capacity, muscle strength and fatigue in sarcoidosis. In this longitudinal study the changes in prevalence of exercise intolerance, reduced muscle strength and fatigue will be established in a two-year follow-up. Also the relation between these physical impairments in time and other clinical parameters, such as QOL, will be established.

Study design: sarcoidosis patients referred to the ild care team of outpatient clinic of the department of Respiratory Medicine of the MUMC and also participated in the baseline study between November 2008 and September 2009 will be included in this longitudinal study. A six-minute walk test and peripheral muscle strength measurements (included in the regular clinical work-up of sarcoidosis patients) will be performed under supervision of a physical therapist at the department of physical therapy of the MUMC. Moreover, the patients will be asked to complete the WHOQOL-bref questionnaire and the Fatigue Assessment Scale. A maximum of 124 patients will be included.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed sarcoidosis according to WASOG/ATS/ERS guidelines

Exclusion Criteria:

* not being able to walk

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Sarcoidosis patients referred to the ild care team of the outpatient clinic of the department of Respiratory Medicine of the Maastricht University Medical Centre (MUMC) a tertiary referral center in the Netherlands will be included in this study
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2009-01; Primary Completion 2009-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Exercise capacity, muscle strength and fatigue in sarcoidosis: a two-year follow-up study | 30 months
  6MWD and muscle strength measurements of arm (isometric strength of the elbow flexors) and leg (isokinetic peak torques of the hamstrings and quadriceps) muscles. Questionnaires: WHOQOL-bref and Fatigue Assessment Scale (FAS).

CONTACTS AND LOCATIONS:
Overall Officials: Rik Marcellis, MSc, Principal Investigator — Maastricht University Medical Center; Marjolein Drent, MD, PhD, Study Chair — Maastricht University Medical Center and University Maastricht; Ton Lenssen, MSc, PhD, Study Director — Maastricht UMC and University of Maastricht
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands

REFERENCES:
- [Result] Marcellis RG, Lenssen AF, Elfferich MD, De Vries J, Kassim S, Foerster K, Drent M. Exercise capacity, muscle strength and fatigue in sarcoidosis. Eur Respir J. 2011 Sep;38(3):628-34. doi: 10.1183/09031936.00117710. Epub 2011 Mar 24. PMID 21436356
- [Derived] Marcellis RG, Lenssen AF, Kleynen S, De Vries J, Drent M. Exercise capacity, muscle strength, and fatigue in sarcoidosis: a follow-up study. Lung. 2013 Jun;191(3):247-56. doi: 10.1007/s00408-013-9456-6. Epub 2013 Apr 5. PMID 23558599
- See also: official site of the Maastricht University Medical Centre — http://www.azm.nl